CLINICAL TRIAL: NCT00789425
Title: A Randomised, Double Blind, Parallel Group, 12-month Comparison of a Standardized Olive Extract With Placebo in Postmenopausal Women With Decreased Bone Mineral Density
Brief Title: Investigating the Effect of Standardized Olive Extract on Bone Turnover Markers in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioActor (Industry)
Responsible Party: Hans van der Saag, BioActor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BA-IMW-POLYPHENOL-001
Record Dates: First submitted 2008-09-30; First posted 2008-11-11 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Osteoporosis; Osteopenia
Keywords: osteoporosis; osteopenia; olive extract; oleuropein
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): a standardized extract of olive polyphenols at 250 mg per day + 1000 mg of calcium per day.
  Interventions: Dietary Supplement: Standardized Extract of Olive Polyphenols
- 2 (Placebo Comparator): Placebo (starch) + 1000 mg of calcium per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Standardized Extract of Olive Polyphenols — Dietary supplement containing 250 mg of a standardized extract of olive polyphenols per day in 1 capsule.
  A supplement with 1000 mg calcium per day will be supplied together with the active treatment.
  Arms: 1
Dietary Supplement: Placebo — Placebo (starch). A supplement with 1000 mg calcium per day will be supplied together with the active treatment.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the intake of a daily dosage of standardized olive extract provides any protection against bone loss.

DETAILED DESCRIPTION:
Apart from estrogen deficiency, the early postmenopausal period is also characterised by an increasing inflammatory and oxidant status, which further contributes to the development of osteoporosis/osteopenia. The link between systemic inflammation and osteoporosis has only been established recently as it was found that higher circulating hsCRP levels are associated with lower bone mineral density in both healthy pre- and postmenopausal women. Furthermore, it was already known for a long time that one of the most important cytokines implicated in the pathogenesis of various metabolic bone diseases, including postmenopausal osteoporosis, is interleukin (IL)-6, which is produced by osteoblasts, monocytes and T-cells.

Olive oil is the principle fat source of the traditional Mediterranean diet, a diet that has been associated with a low incidence of some diseases, including coronary heart disease and osteoporosis. In addition to the main ingredient (ie. oleic acid) extra virgin olive oil also contains phenolic compounds, such as oleuropein- and ligstroside-aglycones and their derivatives. They are formed in olives by enzymatic removal of glucose from the polar parent compound oleuropein-glycoside. A Mediterranean diet rich in olive oil supplies 10 - 20 mg of phenols per day.

The main metabolic attribute of oleuropein is that it exerts both antioxidant and anti-inflammatory activity by lowering the levels of proinflammatory cytokines like IL-1, IL-6 or TNF-alpha. By inhibiting osteoclast activity, this may result in lowering the rate of bone resorption and, at least in part, protect against osteoporosis development.

Formulated as a capsule it is expected that the compliance and tolerability will be improved compared to the liquid administration. The present study is designed to investigate the effect of 250 mg of a standardized extract of olive polyphenols per day on bone loss in postmenopausal women with decreased bone mass (osteopenia) .

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Gender female
* Between 50-70 years of age
* At least 2 years post menopause
* Bone mineral density (BMD) < or equal to -1.5 and > or equal to -2.5 SD% Young Adult
* Patients with stabilised food habits
* Patients able to understand the nature of the study and able to give signed written informed consent.

Exclusion Criteria:

* Patients with any diseases affecting bone tissue e.g. primary hyperparathyroidism.
* Patients during any therapy affecting bone tissue e.g. HRT, corticosteroids.
* Patients with any associated illness of sufficient severity, or clinically relevant abnormalities in the pre-study screening, which in the opinion of the investigator would make them unsuitable for inclusion in the study, e.g. severe heart failure, severe ischaemic heart disease etc.
* Planned hospitalisation (major surgery) during the study.
* Patients who have any known allergy or intolerance to any compound in the test product.
* Patients who are unwilling or unable to comply with the study protocol for any other reason.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Serum levels of Osteocalcin and CTX will be used as bone turnover markers | 0, 3, 6, and 12 months

SECONDARY OUTCOMES:
Bone mineral density as measured by DEXA in lumbar spine and total hip | 0 and 12 months
hs-CRP and IL-6 in serum as inflammation markers | 0, 6, and 12 months
ORAC values in serum as oxidative stress marker | 0, 6, and 12 months
Total cholesterol, HDL-C, LDL-C, triglycerides in serum as CVD-risk markers. | 0, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Filip, MD PhD, Principal Investigator — Institute of Agricultural Medicine
Locations (1):
- Osteoporosis Outpatient of the Institute of Agricultural Medicine, Lublin, Poland

REFERENCES:
- [Derived] Filip R, Possemiers S, Heyerick A, Pinheiro I, Raszewski G, Davicco MJ, Coxam V. Twelve-month consumption of a polyphenol extract from olive (Olea europaea) in a double blind, randomized trial increases serum total osteocalcin levels and improves serum lipid profiles in postmenopausal women with osteopenia. J Nutr Health Aging. 2015 Jan;19(1):77-86. doi: 10.1007/s12603-014-0480-x. PMID 25560820